CLINICAL TRIAL: NCT06913725
Title: An Exploratory Study to Evaluate the Efficacy and Safety of FCN-159 in Patients With Brain Arteriovenous Malformations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Shanghai Fosun Pharmaceutical Industry Development Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hongtao
Record Dates: First submitted 2025-03-18; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Brain Arteriovenous Malformations
Keywords: Brain Arteriovenous Malformation; MEK Inhibitors; Pharmacological Treatment

STUDY DESIGN:
Intervention Model Description: The experimental group will receive the medication. In this study, the patients in the experimental group will be matched 1:1 with control group patients based on factors such as gender, age (±5 years), the anatomical location of the BAVM lesion, and the Spetzler-Martin grade. Patients in the control group will receive no treatment during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open label FCN-159 (Experimental): Participants receive 8mg FCN-159 orally once daily. Participants continue to reveive FCN-159 until disease progression, unacceptable toxicity or other end-of-treatment criteria.
  Interventions: Drug: FCN-159
- No-treatment control (No Intervention): Patients in the control group will undergo conservative observation throughout the study period.

INTERVENTIONS:
Drug: FCN-159 — An investigational oral MEK inhibitor
  Arms: Open label FCN-159

SUMMARY:
A single-center, open-label, non-randomized controlled exploratory study is conducted in the Xuanwu Hospital Capital Medical University to evaluate the efficacy and safety of FCN-159 in patients with brain arteriovenous malformations (BAVM), aiming to overcome the current clinical challenges caused by the lack of available drugs for this disease.

DETAILED DESCRIPTION:
This open-label Phase 2 study will evaluate the efficacy and safety of FCN-159 in participants with BAVM disease who currently deemed unsuitable for surgery, radiotherapy, interventional embolization, or lacking corresponding surgical treatment indications based on investigator judgment. Eligible patients have no prior rupture. This project plans to recruit 10 patients with BAVMs. They are 1：1 divided into FCN-159 group and no-treatment controlled group. It is stratified by gender, age (±5 years), anatomical site of the lesion, Spetzer-Martin grade. FCN-159 will be administered orally and treatment will be continuous, 28 days as a cycle. The major efficacy outcome measure is overall response rate (ORR) assessed by silence MRA. Participants will be evaluated radiologically at 3, 6, 12 treatment cycles after initiation of treatment, and then every 6 treatment cycles and EOT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 60 years.
2. Diagnosis of brain arteriovenous malformation (AVM) confirmed by DSA.
3. Spetzler-Martin grade IV-V
4. No history of rupture of the AVM vessels.
5. No aneurysmal structures that are amenable to interventional embolization.
6. No major surgery within the past 3 months.
7. Able to swallow and retain oral medication, with no significant gastrointestinal abnormalities that could affect drug absorption, such as malabsorption syndrome, bowel obstruction, or extensive gastrointestinal resection.
8. Karnofsky Performance Score ≥ 50%
9. The patient must have adequate organ and bone marrow function, and must not have received blood transfusions or used any supportive medications (such as cytokines or erythropoietin) to elevate white blood cells, platelets, or hemoglobin levels within 7 days prior to screening:

   Absolute neutrophil count ≥ 1.0 × 10^9/L. Hemoglobin ≥ 90 g/L. Platelet count ≥ 100 × 10^9/L. Total serum bilirubin ≤ 1.5 × upper limit of normal (ULN), patients with Gilbert's syndrome may have ≤ 3.0 × ULN.

   Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN.

   Albumin ≥ 3 g/dL. Creatinine < 1.5 × ULN or creatinine clearance ≥ 50 mL/min. Urine protein < 2+; if urine protein ≥ 2+, then 24-hour urine protein quantification must be ≤ 1g.

   Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
10. The patient must voluntarily sign a written informed consent and be able to complete follow-up visits.
11. For patients of reproductive potential: the patient must agree to use an effective contraceptive method, such as combined hormonal contraception, progestin-only contraception with ovulation suppression, intrauterine device (IUD), intrauterine system (IUS), bilateral tubal ligation, partner's vasectomy, or complete abstinence during the treatment period and for at least 90 days after the last dose of study treatment. Male patients should agree to avoid sperm donation for at least 90 days after the last dose of treatment.

Exclusion Criteria:

1. Patients with multiple arteriovenous malformation lesions (excluding segmental lesions such as CAMS syndrome) or extracranial arteriovenous malformation lesions;
2. Diagnosed with Hereditary Hemorrhagic Telangiectasia (HHT), Capillary Malformation-Arteriovenous Malformation syndrome (CM-AVM), PTEN Hamartoma Tumor Syndrome (PHTS), or CLOVES syndrome;
3. Patients who have received one of the following treatments after birth: a. Stereotactic radiation therapy, surgical treatment, or interventional embolization for BAVM; b. Pharmacological treatment for BAVM; c. Participation in other interventional clinical trials for BAVM;
4. History of ruptured bleeding from malformed vascular clusters or other causes of brain hemorrhage, including subarachnoid hemorrhage, before the screening period;
5. Patients with malignant tumors currently or within the past three years, except for non-melanoma skin basal cell carcinoma, in situ breast cancer, or in situ cervical cancer;
6. Unable to undergo MRI scans and/or have contraindications to MRI (e.g., interference with MRI target lesion volume analysis due to prosthetics, braces, etc.);
7. Unable to undergo DSA and/or have contraindications to DSA (e.g., contrast agent allergy, coagulopathy, etc.);
8. Poorly controlled epilepsy;
9. Uncontrolled, unstable hypertension: Repeated measurements showing systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg with antihypertensive treatment;
10. Dysphagia, active gastrointestinal diseases, malabsorption syndrome, or other conditions affecting the absorption of study drugs;
11. Piror or current retinal vein occlusion (RVO), retinal pigment epithelium detachment (RPED), glaucoma, or other significant abnormalities in ophthalmologic examinations;
12. Interstitial lung disease, including clinically significant radiation pneumonitis;
13. Cardiac function or comorbidities that meet one of the following conditions: a. Three 12-lead ECG measurements conducted during the screening period at the study center, with an average QTcF >470 ms calculated using the QTcF formula for the instruments employed; presence of risk factors for QTcF prolongation, such as uncorrectable hypokalemia, inherited long QT syndrome, or taking drugs known to prolong QTcF (mainly Class Ia, Ic, III antiarrhythmic drugs). New York Heart Association (NYHA) functional classification ≥3 congestive heart failure; c. Clinically significant arrhythmias, including but not limited to complete left bundle branch block; d. Documented, clinically significant coronary artery disease, cardiomyopathy, or severe valvular heart disease; e. Echocardiogram showing left ventricular ejection fraction (LVEF) <50%; f. Bradycardia with a heart rate <50 beats per minute;
14. Family history of sudden cardiac death before the age of 50 in a first-degree relative;
15. Active bacterial, fungal, or viral infections, including active hepatitis B (positive hepatitis B surface antigen and hepatitis B virus DNA >1000 IU/ml, or meeting the study center's criteria for active hepatitis B infection), hepatitis C (positive hepatitis C virus RNA), or HIV infection (HIV positive);
16. Pregnant or breastfeeding women;
17. Known allergy to the study drug, other MEK1/2 inhibitors, or excipients;
18. Any other factors determined by the investigator that may lead to forced discontinuation of the trial, such as severe diseases (including psychiatric disorders) requiring concomitant treatment, significant laboratory abnormalities, family or social factors that may affect the subject's safety or data collection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by Silence-MRA | 1 year

SECONDARY OUTCOMES:
DSA-assessed ORR (Objective Response Rate). | 1 year
Changes in lesion volume at 3 months on Silence-MRA | 3 months
Changes in lesion volume at 6 months on Silence-MRA | 6 months
Changes in lesion volume at 12 months on Silence-MRA | 12 months
Changes in lesion volume at 12 months assessed by DSA | 12 months
Changes in blood flow velocity of feeding arteries assessed by MRI | 12 months
Changes in venous drainage flow velocity assessed by MRI | 12 months
Changes in microhemorrhage around the malformation assessed by MRI | 12 months
Changes in iron deposition around the malformation assessed by MRI. | 12 months
Changes in cerebral perfusion assessed by MRI | 12 months
Intracranial hemorrhage event. | 12 months
The occurrence of epilepsy events. | 12 months
Change in mRS score compared to baseline | 12 months
The types of adverse events occurring during treatment (TEAEs） | 12 months
The frequency of adverse events occurring during treatment (TEAEs) | 12 months

OTHER OUTCOMES:
Maximum Plasma Concentration [Cmax] | 3 months, 6 months, 12 months
Area under the plasma concentration versus time curve (AUC) | 3 months, 6 months, 12months

CONTACTS AND LOCATIONS:
Locations (1):
- the Department of Neurosurgery, China International Neuroscience Institute, Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
From 6 months post analysis and article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept Department of Neurosurgery, Xuanwu Hospital, Capital Medical University conditions for access:
  * Individual participant data that underlie the results reported in this article after de- identification
  * Trial protocol,Statistical Analysis Plan,PICF The Sponsor-Investigator will be the long-term custodian after the archive period has finished.
Supporting Information: Study Protocol
Time Frame: Available from 6 months following analysis and article publication
Access Criteria: Future researchers must be from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept Department of Neurosurgery, Xuanwu Hospital, Capital Medical University's conditions for access
URL: https://www.xwhosp.com.cn/